CLINICAL TRIAL: NCT05076136
Title: Comparison of Regional Manual Therapy and Standard Physical Therapy Intervention in Females With Sacroiliac Joint Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCRS/20/1017
Record Dates: First submitted 2021-09-29; First posted 2021-10-13 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Sacroiliac; Sprain (Strain)
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regional treatment (Experimental): Group A was given regional treatment with baseline treatment protocol
  Interventions: Other: Regional treatment
- Standard physiotherapy treatment (Active Comparator): Group B was given standard physiotherapy treatment with baseline protocol
  Interventions: Other: Standard physiotherapy treatment

INTERVENTIONS:
Other: Regional treatment — In reginal treatment patients were given physiotherapy exercises and manual therapies on hip joint as well as on surrounding areas of hip joint such as lumber area and sacroiliac joint.
  Arms: Regional treatment
Other: Standard physiotherapy treatment — In this treatment patients were given just hip joint mobilizations and quadriceps and hamstrings stretching.
  Arms: Standard physiotherapy treatment

SUMMARY:
The SIJ has long been considered an important source of low back pain because of the empirical ﬁnding that treatment targeting the SIJ can relieve pain.This study was be a Randomized Clinical Trail conducted at Riphah Rehabilitation Centre Lahore. The study was be completed within the time duration of Six months. Purposive sampling technique was be used. Sample size is calculated by using the G power 3.1. The sample size of 64 patients was be taken in this study to find the comparison of regional manual therapy and standard physiotherapy intervention in females with sacroiliac joint pain. Patients was be divided into two groups.. Patients was be divided into two groups. Group A was be treated with regional manual therapy. In regional manual therapy patients was be given mobilization to lumber region and SIJ, pelvic floor exercises and core strengthening exercises and Group B was be treated with standard physiotherapy in which patients was be given SIJ mobilization and Straight leg raise. Both groups was receive transcutaneous electrical nerve stimulator and heating pad as a common treatment protocol. Numeric pain rating scale (NPRS) and oswestry low back disability questionnaire was be used as Data collecting tools. Two session of treatment per week for eight weeks was be given. Data was be analyzed on SPSS 21.

ELIGIBILITY:
Inclusion Criteria:

* Females with sacroiliac joint pain
* Age: 20 to 50 years

Exclusion Criteria:

* Patients withany red flag signs i.etumor, fracture, metabolic diseases, rheumatoid arthritis, prolonged history of steroids use, etc.
* Females with sciatica
* Females with radiating pain

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2019-11-24 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
NPRS | Eight week
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.
Oswestry low back disability questionnaire | Eight week
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools

CONTACTS AND LOCATIONS:
Overall Officials: Tasneem Shahzadi, Mphil, Study Chair — Riphah international university Lahore
Locations (1):
- Bajwa hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forst SL, Wheeler MT, Fortin JD, Vilensky JA. The sacroiliac joint: anatomy, physiology and clinical significance. Pain Physician. 2006 Jan;9(1):61-7. PMID 16700283
- [Background] 5. Merskey H, Bogduk N. Classiﬁcation of Chronic Pain:Descriptions of Chronic Pain Syndromes and Deﬁnitions of Pain Terms. 2nd ed. Seattle, WA: IASP Press; 1994.
- [Background] 7. Solonen KA: The sacroiliac joint in the light of anatomical, roentgenological and clinical studies. Acta Orthop Scand 1957;27(suppl):1-127 Fortin JD, Dwyer AP, West S, et al: Sacroiliac joint: pain referral maps upon applying a newinjection/arthrography technique: part 1, asymptomatic volunteers. Spine 1994; 19(13):1475-1482